CLINICAL TRIAL: NCT01219764
Title: A Randomized Trial of Standard vs Half Dose Rabeprazole, Clarithromycin, Metronidazole and Amoxicillin in the Treatment of Helicobacter Pylori Infection
Brief Title: A Trial of Standard vs Half Dose Rabeprazole, Clarithromycin, Metronidazole and Amoxicillin in the Treatment of Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Ala'a Sharara, Professor of Medicine, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM.AS1.25
Record Dates: First submitted 2010-05-19; First posted 2010-10-13 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Helicobacter Infections
Keywords: Helicobacter pylori infection; quadruple therapy; Amoxicillin; Metronidazole; Clarithromycin; Rabeprazole
MeSH Terms: conditions — Helicobacter Infections | interventions — Rabeprazole; Metronidazole; Clarithromycin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Full Dose (Active Comparator): Full dose of Rabeprazole (20mg), metronidazole (500mg), Clarithromycin (500mg) and Amoxicillin (1000mg) twice daily for a period of 7 days.
  Interventions: Drug: Rabeprazole, metronidazole, Clarithromycin, Amoxicillin
- Half dose (Experimental): Rabeprazole (10mg), metronidazole (250mg), Clarithromycin (250mg) and Amoxicillin (500mg) twice daily for a period of 7 days.
  Interventions: Drug: Rabeprazole, metronidazole, Clarithromycin, Amoxicillin

INTERVENTIONS:
Drug: Rabeprazole, metronidazole, Clarithromycin, Amoxicillin — Full dose arm:Rabeprazole (20mg), metronidazole (500mg), Clarithromycin (500mg) and Amoxicillin (1000mg) twice daily for a period of 7 days.
  Half dose arm: Rabeprazole (10mg), metronidazole (250mg), Clarithromycin (250mg) and Amoxicillin (500mg) twice daily for a period of 7 days.
  Other Names: Rabeprazole: Pariet; Metronidazole: Flagyl; Clarithromycin: Klacid; Amoxicillin: Amoxil

SUMMARY:
The proposed study will test the hypothesis that H. pylori can be eradicated successfully (>85%) using half-or full-dose "concomitant" non-bismuth quadruple therapy regimen: rabeprazole, amoxicillin, clarithromycin and metronidazole twice daily for 7 days in patients with peptic ulcers and H. pylori related gastritis.

Two hundred patients from the outpatient department and the endoscopy unit at AUBMC will be enrolled in this open-label trial. Patients with positive CLO tests or urea breath tests, documenting H.pylori infection, will be randomized into one of two groups: Full dose or half dose the concomitant regimen, with 100 patients in each group. Compliance and side effects will be assessed, and a urea breath test will be done for all patients after 4 weeks of therapy completion to evaluate eradication rates. Success of therapy will be evaluated according to intent-to treat and per-protocol analyses.

DETAILED DESCRIPTION:
Infection with H. pylori has been linked with chronic active gastritis, peptic ulcer disease, adenocarcinoma and Non-Hodgkin's lymphoma of the stomach. Eradication of this organism has been recommended for patients with peptic ulcer disease, low-grade gastric mucosa-associated lymphoid tissue lymphoma, atrophic gastritis, unexplained iron deficiency anemia, chronic idiopathic thrombocytopenic purpura, as well as first-degree relatives of gastric cancer patients.

Guidelines still recommend using triple therapy regimen of PPI, clarithromycin and amoxicillin/metronidazole twice daily for 7 to 14 days. Over the years, it has become clear that the first-line triple therapy is loosing efficacy worldwide with PP and ITT eradication rates inferior to 80%. Antimicrobial resistance plays an important role in some of these failures.

Major H. pylori study groups in the world have agreed that alternative treatment regimens are urgently needed. So far, 2 alternative treatment regimens have shown superiority over the first-line treatment protocols: the sequential therapy consisting of a combination of amoxicillin and a PPI twice a day for 5 days followed by another 5 days of the PPI plus clarithromycin and tinidazole/metronidazole, and the concomitant non-bismuth quadruple regimen consisting of PPI, clarithromycin, metronidazole, and amoxicillin twice daily.

The proposed study will test the hypothesis that H. pylori can be eradicated successfully (>85%) using half-or full-dose "concomitant" non-bismuth quadruple therapy regimen: rabeprazole, amoxicillin, clarithromycin and metronidazole twice daily for 7 days in patients with peptic ulcers and H. pylori related gastritis.

Two hundred patients from the outpatient department and the endoscopy unit at AUBMC will be enrolled in this open-label trial. Patients with positive CLO tests or urea breath tests, documenting H.pylori infection, will be randomized into one of two groups: Full dose or half dose the concomitant regimen, with 100 patients in each group. Compliance and side effects will be assessed, and a urea breath test will be done for all patients after 4 weeks of therapy completion to evaluate eradication rates. Success of therapy will be evaluated according to intent-to treat and per-protocol analyses.

ELIGIBILITY:
Inclusion Criteria:

* documented H.pylori infection by a CLO test or a Urea Breath Test
* sign the informed consent

Exclusion Criteria:

* Age under 18 or older than 80 years
* Allergies to any of the drugs used
* Recent antibiotic therapy (within 2 weeks of enrolment)
* Severe ulcers or bleeding
* Gastric perforation or obstruction
* Previous gastrectomy
* Gastric cancer
* Pregnancy or lactation
* Prior eradication therapy for H. pylori
* Severe concomitant disease or condition making the treatment unlikely to be effective i.e. alcoholism, drug addiction, and history of poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with negative urea breath test post treatment | 30 days post treatment completion
  30 days post treatment completion, patients will do a Urea Breath Test (a test that is regularly used to check for H. Pylori infection in the stomach) to check whether H. Pylori has been eradicated from the stomach or not.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | during the 7 days of the treatment
  we will check for nausea, vomiting, metallic taste, diarrhea, and abdominal pain during the 7 days of the treatment period in each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ala' I Sharara, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut - Medical Center, Beirut, Lebanon